CLINICAL TRIAL: NCT04881617
Title: Establishing Evidence-based Treatment for Speech and Language in Primary Progressive Aphasia
Brief Title: Treatment for Speech and Language in Primary Progressive Aphasia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DC016291 (NIH); R01DC016291 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Primary Progressive Aphasia; Semantic Dementia; Semantic Memory Disorder; Logopenic Progressive Aphasia; Nonfluent Aphasia, Progressive; Aphasia; Aphasia, Progressive
MeSH Terms: conditions — Aphasia, Primary Progressive; Frontotemporal Dementia; Memory Disorders; Primary Progressive Nonfluent Aphasia; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lexical Retrieval Treatment (Experimental)
  Interventions: Behavioral: Lexical Retrieval Training (LRT)
- Script Training (Experimental)
  Interventions: Behavioral: Video-Implemented Script Training for Aphasia (VISTA)

INTERVENTIONS:
Behavioral: Lexical Retrieval Training (LRT) — In person or via teletherapy: Participants work on producing spoken and written names of personally relevant target items using a self-cueing hierarchy. Treatment focuses on the use of strategies that capitalize on spared cognitive-linguistic abilities to support word retrieval. The participant completes two (one hour each) sessions per week with a clinician plus daily home practice exercises.
  Arms: Lexical Retrieval Treatment
Behavioral: Video-Implemented Script Training for Aphasia (VISTA) — In person or via teletherapy: Participants work on producing personally relevant scripts of 4-6 sentences in length. Length and complexity of scripts are individually tailored. The participant completes 30 minutes per day of home practice, during which they speak in unison with a video/audio model of a healthy speaker clearly articulating the scripts. Biweekly (one hour each) sessions with a clinician target clear and accurate script production, script memorization, and conversational usage of scripts.
  Arms: Script Training

SUMMARY:
Primary progressive aphasia (PPA) is a progressive neurological disorder that causes a gradual decline in communication ability as a result of selective neurodegeneration of speech and language networks in the brain. PPA is a devastating condition affecting adults as young as their 40's or 50's, depriving them of the ability to communicate and function in society. There has been significant progress in discovering the neurobiological mechanisms that underlie PPA and in identifying its clinical phenotypes. With these advances, we are poised to investigate behavioral treatments that are grounded in modern cognitive and neuroanatomical concepts. Research documenting the efficacy of speech-language treatment for PPA is emerging, but limited. Systematic research is needed to establish best clinical practices in this unique patient population for whom pharmacological treatment remains elusive. The long-term objectives of this project are to provide evidence-based treatment methods addressing the speech and language deficits in PPA and to determine the neural predictors of responsiveness to intervention. The study has three main goals that build on the findings of our previous work: 1) to examine the utility of treatments designed to facilitate significant, generalized and lasting improvement of speech-language function in PPA, 2) to determine whether treatment alters the trajectory of decline in PPA by comparing performance on primary outcome measures in treated versus untreated participants after a one-year interval, and 3) to identify imaging predictors (gray matter, white matter, and functional connectivity measures) of responsiveness to behavioral intervention in individuals with PPA. In order to accomplish these aims, we will enroll 60 individuals with PPA, who will undergo a comprehensive multidisciplinary evaluation and neuroimaging. Subsequently, participants will be enrolled in treatment designed to promote lasting and generalized improvement of communicative function in core speech-language domains. Participants will be followed for up to one-year post-treatment in order to determine long-term effects of rehabilitation, and their performance will be compared with a historical cohort of untreated PPA patients. This ambitious study and the necessary recruitment will be possible due to an ongoing collaboration with the UCSF Memory and Aging Center, a leading institution in the field of PPA research. The study will broaden the evidence base supporting the efficacy of speech-language intervention in PPA and will provide novel evidence regarding neural predictors of treatment outcomes, with the potential to inform clinical decision-making and improve clinical care for individuals with this debilitating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for Primary Progressive Aphasia (PPA; Gorno-Tempini et al., 2011)
* Score of 15 or higher on the Mini-Mental State Examination

Exclusion Criteria:

* Other neurological or psychiatric diagnosis that may contribute to cognitive-linguistic deficits
* Significant, uncorrected visual or hearing impairment that would interfere with participation
* Score of less than 15 on the Mini-Mental State Examination
* Prominent initial non-speech-language impairment (cognitive, behavioral, motoric)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in spoken naming of target items | change from pre-treatment to post-treatment (approximately 8-12 weeks after treatment onset) and follow-ups at 3 months post-treatment, 6 months post-treatment, and 12 months post-treatment
  Change in percent correctly named trained/untrained pictures
Change in script production accuracy | change from pre-treatment to post-treatment (approximately 6 weeks after treatment onset) and follow-ups at 3 months post-treatment, 6 months post-treatment, and 12 months post-treatment
  Change in percent correct intelligible, scripted words for trained/untrained scripts

SECONDARY OUTCOMES:
Change on Western Aphasia Battery, Revised | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment, 6 months post-treatment, and 12 months post-treatment
  change on standardized aphasia assessment
Change on Boston Naming Test | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment, 6 months post-treatment, and 12 months post-treatment
  change on standardized word retrieval assessment
Change on Northwestern Assessment of Verbs and Sentences | change from pre-treatment to post-treatment (approximately 6-12 weeks after treatment onset) and follow-ups at 3 months post-treatment, 6 months post-treatment, and 12 months post-treatment
  change on standardized assessment of verb and sentence processing in aphasia

OTHER OUTCOMES:
Post-treatment Communication Survey | post-treatment (approximately 6-12 weeks after treatment onset)
  survey characterizing perceived response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maya L Henry, PhD, Principal Investigator — University of Texas at Austin
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - University of Texas, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry ML, Hubbard HI, Grasso SM, Mandelli ML, Wilson SM, Sathishkumar MT, Fridriksson J, Daigle W, Boxer AL, Miller BL, Gorno-Tempini ML. Retraining speech production and fluency in non-fluent/agrammatic primary progressive aphasia. Brain. 2018 Jun 1;141(6):1799-1814. doi: 10.1093/brain/awy101. PMID 29718131
- [Background] Henry ML, Hubbard HI, Grasso SM, Dial HR, Beeson PM, Miller BL, Gorno-Tempini ML. Treatment for Word Retrieval in Semantic and Logopenic Variants of Primary Progressive Aphasia: Immediate and Long-Term Outcomes. J Speech Lang Hear Res. 2019 Aug 15;62(8):2723-2749. doi: 10.1044/2018_JSLHR-L-18-0144. Epub 2019 Aug 7. PMID 31390290
- [Background] Dial HR, Hinshelwood HA, Grasso SM, Hubbard HI, Gorno-Tempini ML, Henry ML. Investigating the utility of teletherapy in individuals with primary progressive aphasia. Clin Interv Aging. 2019 Feb 25;14:453-471. doi: 10.2147/CIA.S178878. eCollection 2019. PMID 30880927
- See also: University of Texas Aphasia Research and Treatment Lab — https://slhs.utexas.edu/research/aphasia-research-treatment-lab
- See also: UCSF Language Neurobiology Lab — https://albalab.ucsf.edu